CLINICAL TRIAL: NCT05192889
Title: RAVEN: A Phase I/II Trial Treating Relapsed Acute Lymphoblastic Leukemia With Venetoclax and Navitoclax
Brief Title: Trial Treating Relapsed Acute Lymphoblastic Leukemia With Venetoclax and Navitoclax
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RAVEN; NCI-2022-00304 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-01-11; First posted 2022-01-14 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Refractory Acute Lymphoblastic Leukemia; Relapsed Acute Lymphoblastic Leukemia
Keywords: Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia; Children; Young Adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; navitoclax; Dexamethasone; Calcium Dobesilate; Vincristine; calaspargase pegol; Dasatinib; Cytarabine; blinatumomab; Methotrexate; Mercaptopurine; Cyclophosphamide; Etoposide; Leucovorin; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Radiation

STUDY DESIGN:
Intervention Model Description: All eligible patients receive a common first block of therapy and therapy in the 2nd block being determined by CD19 expression on leukemic blasts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Block 1 (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Navitoclax, Dexamethasone, Vincristine, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Dasatinib, Leucovorin, Intrathecal (IT) MHA (methotrexate/hydrocortisone/cytarabine)
  Interventions: Drug: Venetoclax; Drug: Navitoclax; Drug: Dexamethasone; Drug: Vincristine; Drug: Calaspargase Pegol; Drug: Dasatinib; Drug: Leucovorin; Drug: Intrathecal Triples; Drug: Pegaspargase; Drug: Erwinia asparaginase
- Block 2 (Experimental): Block 2a Therapy:
  Patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Navitoclax, Dexamethasone, Cytarabine, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Dasatinib, IT MHA, Radiation
  Block 2b Therapy:
  Patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Blinatumomab, Dexamethasone, Dasatinib, IT MHA
  Following Block 2 of therapy, late (≥36 months from diagnosis) first relapse B-ALL who are MRD negative after Block 1 will continue chemotherapy using adapted R3 intensification, interim, and continuation therapies.
  Patients receive intervention according to the Detailed Description section with the following:
  Methotrexate, Mercaptopurine, IT MHA, Leucovorin, Dexamethasone, Vincristine, Cyclophosphamide, Etoposide, Cytarabine, Dasatinib, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Radiation
  Interventions: Drug: Venetoclax; Drug: Navitoclax; Drug: Dexamethasone; Drug: Vincristine; Drug: Calaspargase Pegol; Drug: Dasatinib; Drug: Cytarabine; Biological: Blinatumomab; Drug: Methotrexate; Drug: Mercaptopurine; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Leucovorin; Drug: Intrathecal Triples; Drug: Pegaspargase; Drug: Erwinia asparaginase; Radiation: Radiation

INTERVENTIONS:
Drug: Venetoclax — Given oral (PO).
  Other Names: Venclextra®; ABT-199
Drug: Navitoclax — Given oral (PO).
  Other Names: ABT-263
Drug: Dexamethasone — Given orally (PO) or intravenously (IV).
  Other Names: Decadron®; Hexadrol®; Dexameth®
Drug: Vincristine — Given intravenously (IV).
  Other Names: Vincristine sulfate; Oncovin®
Drug: Calaspargase Pegol — Given intravenously (IV).
  Other Names: Asparlas
Drug: Dasatinib — Given oral (PO).
  Other Names: Sprycel®
Drug: Cytarabine — Given intravenously (IV) or Intrathecal (IT).
  Other Names: Ara-C; Cytosar-U®
  Arms: Block 2
Biological: Blinatumomab — Given intravenously (IV).
  Other Names: Blincyto®
  Arms: Block 2
Drug: Methotrexate — Given intravenously (IV), oral (PO), or Intrathecal (IT).
  Other Names: MTX; Trexall®; amethopterin
  Arms: Block 2
Drug: Mercaptopurine — Given oral (PO).
  Other Names: 6-MP; Purinethol®
  Arms: Block 2
Drug: Cyclophosphamide — Given intravenously (IV).
  Other Names: Cytoxan®
  Arms: Block 2
Drug: Etoposide — Given intravenously (IV).
  Other Names: VP-16; Vepesid®
  Arms: Block 2
Drug: Leucovorin — Given oral (PO) or intravenously (IV).
  Other Names: Folinic acid
Drug: Intrathecal Triples — Given Intrathecal (IT).
  Other Names: ITMHA; methotrexate/hydrocortisone/cytarabine
Drug: Pegaspargase — May be used in place of Calaspargase Pegol where available. Given intravenously (IV) or intramuscularly (IM).
  Other Names: Oncaspar®; PEG-asparaginase; PEG-L-asparaginase
Drug: Erwinia asparaginase — To be used in case of hypersensitivity or intolerance to Calaspargase Pegol or Pegaspargase. Given intravenously (IV) or intramuscularly (IM).
  Other Names: Erwinase®
Radiation: Radiation — See detailed description section.
  Other Names: Irradiation
  Arms: Block 2

SUMMARY:
This is a phase I/II clinical trial evaluating the activity of combination chemotherapy with venetoclax and navitoclax in children with relapsed or refractory acute lymphoblastic leukemia or lymphoma (rALL) and assessing the combination dose of venetoclax combinations with either blinatumomab for CD19-positive patients or navitoclax and high-dose cytarabine for CD19-negative patients.

Primary Objectives

* To compare Minimal Residual Disease (MRD)-negative CR/CRi rate in children with relapsed or refractory acute lymphoblastic leukemia or lymphoma (rALL) following Block 1 therapy with venetoclax and navitoclax based reinduction to historical controls.
* To identify the recommended phase 2 combination dose (RP2D) of venetoclax based consolidation in novel combinations with a) high-dose cytarabine and navitoclax or b) blinatumomab.

Secondary Objectives

* To estimate the tolerability and activity of venetoclax based consolidation in novel combinations with a) high-dose cytarabine and navitoclax or b) blinatumomab.
* To describe event-free and overall survival in patients treated with this regimen.

Exploratory Objectives

* To evaluate MRD-negative CR/CRi rates in each prespecified groups: late first relapse B-ALL; early first relapse and second or greater relapse B-ALL; and relapsed T-ALL.
* To identify drug sensitivity patterns in patient samples prior to and after receiving combination therapy and evaluate mechanisms of disease resistance/ escape.
* To explore immune subsets during and after this regimen.
* Evaluate response to therapy in rare relapse patient subsets.
* Explore breakthrough infections in children and young adults with relapsed or refractory ALL

DETAILED DESCRIPTION:
This is a non-randomized phase I/II clinical trial. In Block I, all patients receiving common therapy evaluating the activity of combination chemotherapy with venetoclax and navitoclax in children with relapsed or refractory acute lymphoblastic leukemia or lymphoma (rALL).

In Block 2, a phase 1 rolling six design and phase 2 extension will be used to assess the combination dose of venetoclax combinations with either blinatumomab for CD19-positive patients or navitoclax and high-dose cytarabine for CD19-negative patients. One to six participants can be concurrently enrolled onto a dose level, depending on the number of participants enrolled at the current dose level, the number of participants who have experienced a dose/combination limiting toxicity (DLT) at the current dose level, and the number of participants entered but with tolerability data pending. Dose de-escalation will occur if 2 patients at a dose level experience a targeted toxicity. If 6 patients complete a therapy block and experience 0-1 DLT, that dose will be considered the recommended phase 2 dose (RP2D). New enrollment on an arm (2a/2b) will be paused if further enrollment would result in more than 6 patients being treated on that arm before the RP2D is identified.

The primary outcome assessment will be a bone marrow with MRD testing on Day 29 of Block 1 therapy. Following that assessment, patients should continue with protocol therapy including either Block 2A (which includes high-dose cytarabine with venetoclax and navitoclax) for patients with CD19 negative leukemia, those with isolated extramedullary relapse, or whose treating physician determines that blinatumomab therapy is not in the patient's best interest; or Block 2B for patients with leukemia which is CD19 positive. Following recovery from Block 2 therapy, all patients except those with late first relapse of B-ALL (≥ 36 months from diagnosis) who are MRD-negative at <0.01% after Block 1 therapy are off therapy. Further therapy for these patients is at the treating physician's discretion. Patients with late first relapse B-ALL relapse and who are MRD negative will proceed with intensification, interim continuation, and continuation therapy. Patients with Down's Syndrome with CD19 negative leukemia will be off therapy after Block 1 as they are ineligible for Block 2A. Patients in exploratory cohorts I and N who are late first relapse B-ALL and who are MRD-negative after Block 1 therapy may continue on protocol therapy after Block 2 or receive alternative therapy at their treating physician's discretion. Patients in exploratory cohort M and O are off therapy after Block 2.

Intervention:

Block 1 Therapy:

* Venetoclax 120mg/m^2 (max 200mg) PO, day 1; 240mg/m^2/dose (max 400mg) PO, 21 doses, days 2-22
* Navitoclax 25mg PO (for patients 20 - <45kg) OR 50mg PO (for patients >=45kg), days 3-22
* Dexamethasone 5mg/m^2/dose BID PO/IV, days 1-7 and 15-22
* Vincristine 1.5mg/m^2/dose (max 2mg) IV, days 1, 8, 15, and 22
* Calaspargase pegol 2500units/m^2/dose IV, day 2
* Dasatinib 80mg/m^2/day (max 140mg) PO, days 1-28 for ABL-class fusions and non-ETP T-ALL
* IT MHA: Intrathecal (IT) MHA (methotrexate 12 mg/hydrocortisone 24mg/cytarabine 36mg), days -7 to 1. Continue intrathecal chemotherapy weekly until negative x 2.
* Leucovorin 5mg/m2 (max 5mg) PO or IV (24 and 30 hours after each LP).

Calaspargase may be replaced by alternative forms of asparaginase due to local practice or prior allergy. If pegaspargase is used, two doses (on days 2 and 15) of 2500units/ m^2 replace the single day 2 dose of calaspargase. For patients in exploratory cohort N, asparaginase will be omitted. For patients in exploratory cohort O, the Day 15 dose of pegaspargase may be omitted and the Day 2 dose may be capped at 2000units/m2 with a maximum dose of 3750 units.

Testicular Radiation: Patients with persistent testicular involvement by leukemia at the end of Block 1 may continue on study and may receive testicular radiation during Block 2 therapy.

Block 2a - For patients with ≥ 5% of leukemic blasts which do not have detectable CD19 on their surface, those with isolated extramedullary relapse, or whose physician determines this therapy arm is in their patient's best interest. Patients with Down Syndrome are not eligible for Block 2a therapy. Patients in exploratory cohort O are not eligible for the phase I/dose de-escalation phase of the study but may enroll on block 2 therapy after the dose has been established.:

* Venetoclax 240mg/m^2 (max 400mg) PO, days 1-7
* Navitoclax 25mg (20-<45kg) OR 50mg (>=45kg) PO, days 1-7
* Dexamethasone 3mg/m^2/dose PO/IV BID, days 1-5
* Calaspargase pegol 1000units/m^2 IV, day 3
* Dasatinib 80mg/m2/day (max 140mg) PO, days 1-28 for ABL-class fusion and non-ETP T-ALL/ALLy
* IT MHA: Methotrexate 12 mg IT, Hydrocortisone 24mg IT, Cytarabine 36mg IT, one dose with end of cycle bone marrow assessment
* Cytarabine dosing during phase I portion for Block 2a:

  * Dose level 1: 3000mg/m^2/dose every 12hours(h) IV infusion over 3 hours, days 1-2
  * Dose level 0: 1500mg/m^2/dose every 12h IV infusion over 3 hours, days 1-2
  * Dose level -1: 1000mg/m^2/dose every 12h IV infusion over 3 hours, day 1

Calaspargase may be replaced by alternative forms of asparaginase. For patients in exploratory cohort N, asparaginase will be omitted.

Block 2b Therapy: For patients with >95% of leukemic blasts with detectable CD19 on their surface. Patients with isolated extramedullary relapse are ineligible for Block 2b therapy. Patients in exploratory cohort O are not eligible for the phase I/ dose de-escalation phase of the study but may enroll on block 2 therapy after the dose has been established.

* Blinatumomab; for patients with end of Block 1 MRD >5%, 5mcg/m^2/day (max 9mcg/day; patients weighing ≥45kg receive 9mcg/day fixed dose) IV, days 1-7
* Blinatumomab; for patients with end of Block 1 MRD >5%, 15mcg/m^2/day (max 28mcg/day; patients weighing ≥45kg receive 28mcg/day fixed dose) IV, days 8-28
* Blinatumomab; for patients with end of Block 1 MRD ≤5%, 15mcg/m^2/day (max 28mcg/day; patients weighing ≥45kg receive 28mcg/day fixed dose) IV, days 1-28,
* Dexamethasone 10mg/m^2 (max 20mg) 30-60 minutes prior to day 1 blinatumomab, PO/IV, days 1, 8 (For patients who start blinatumomab at 5mcg/m2/day, an additional dose of dexamethasone will be given on day 8 30-60 minutes prior to dose increase. For patients whose blinatumomab is interrupted for more than 4 hours for any reason, an additional dose of dexamethasone will be given prior to restarting blinatumomab.)
* Dasatinib 80mg/m^2/day (max 140mg) PO, days 1-28 for ABL-class fusions
* IT MHA: Methotrexate 12 mg IT, Hydrocortisone 24mg IT, Cytarabine 36mg IT, day 29 with end of cycle bone marrow
* Venetoclax dosing during phase I portion for Block 2b:

  * Dose level 1: 240mg/m^2 (max 400 mg) PO, days 8-28
  * Dose level 0: 240mg/m^2 (max 400 mg) PO, days 8-21
  * Dose level -1: 240mg/m^2 (max 400 mg) PO, days 8-14

Intensification Therapy - For late first relapse B-ALL and MRD<0.01% after Block 1 only. Patients in exploratory cohort O are excluded.:

* High Dose (HD) Methotrexate 5000mg/m^2/dose IV: 500mg/m^2 over 60 minutes then 4500mg/m^2 over 23 hours; or targeted 65 microM, day 1 and 15
* Mercaptopurine 50mg/m^2/dose PO daily, days 1-28
* IT MHA: Methotrexate 12 mg IT, Hydrocortisone 24mg IT, Cytarabine 36mg IT, D15
* Leucovorin 15mg/m2/dose PO/IV every 6 hours (start 42 hours after HD-MTX begins) D2 and 16 (at least 3 doses).

Interim Continuation Therapy 1 and 2 (8 weeks each) - For late first relapse B-ALL and MRD<0.01% after Block 1 only:

* Dexamethasone 3mg/m^2/dose BID PO/IV, days 1-5
* Vincristine1.5mg/m^2(max 2mg) IV, day 1
* Mercaptopurine 75mg/m^2/dose PO daily or 60mg/m2/day for patients with known heterozygous inactivating mutations of TPMT or NUDT15, days 1-49
* Methotrexate 20mg/m^2/dose PO/IV, days 8, 15, 29, 36
* High Dose (HD)-Methotrexate 5000mg/m^2/dose IV: 500mg/m2 over 60 minutes then 4500mg/m^2 over 23 hours; or targeted 65 microM, day 22
* Leucovorin 15mg/m^2/dose PO/IV every 6 hours: Start 42 hours after HD-MTX, days 24 and 25 (at least 3 doses)
* Cyclophosphamide 300mg/m^2/dose IV over 15-30 minutes, days 43 and 50
* Etoposide 150mg/m^2/dose IV over 1-2 hours, days 43 and 50
* Cytarabine 50mg/m^2/dose IV over 1-30 minutes, days 44-47 and 51-54
* Dasatinib 80mg/m^2/day PO (Max 140mg), days 1-56 for ABL-class fusions
* IT MHA: Methotrexate 12 mg IT, Hydrocortisone 24mg IT, Cytarabine 36mg IT, days 22 and 43

Following recovery from Interim Continuation therapy 1, patients will repeat Block 2 therapy according to their initial Block assignment (2A for CD19-negative, 2B for CD19-positive) and receive a second cycle of interim continuation. Patients will not receive venetoclax or navitoclax during this repeated Block 2 cycle. Following recovery from Interim Continuation 2, patients will proceed to Continuation therapy.

Continuation Therapy - For late first relapse B-ALL and MRD <0.01% after Block 1 only. Continuation cycles last 8 weeks (56 days) each. Continuation therapy continues until 2 years from the start of protocol therapy.:

* Dexamethasone 6mg/m^2/dose BID PO/IV, days 1-5, 29-33
* Vincristine 1.5mg/m^2 (max 2mg) IV, day 1 and 29
* Mercaptopurine 75mg/m^2/dose PO daily or 60mg/m^2/day for patients with known heterozygous inactivating mutations of TPMT or NUDT15 days 1-56
* Methotrexate 20mg/m^2/dose PO/IV days 8, 15, 22, 36, 43 and 50
* Dasatinib 80mg/m^2/day PO (Max 140mg) days 1-56 for ABL-class fusions
* IT MHA: Methotrexate 12 mg IT, Hydrocortisone 24mg IT, Cytarabine 36mg IT day 1 and 29 (patients with CNS2 or traumatic lumbar puncture with blasts present at the time of relapse will receive day 1 and 29 IT MHA for the first year of continuation therapy. Following this, patients will receive IT MHA on day 1 of each cycle until the completion of therapy. Patients with CNS3 disease at relapse will receive day 1 and 29 IT MHA during cycles 1 and 2 of continuation and then proceed to chemoradiation.)

Chemoradiation for those with CNS3 disease at relapse (late first relapse [≥36 months from diagnosis] B-ALL and MRD<0.01% after Block 1 only):

Patients with CNS3 disease at relapse will receive 18Gy cranial irradiation after Cycle 2 of Continuation Therapy. Patients will not receive additional intrathecal chemotherapy following irradiation. Chemoradiation lasts 21 days.

* Dexamethasone 6mg/m2/dose BID PO/IV days 1-5 and 15-19
* Vincristine 1.5mg/m^2 (max 2mg) IV days 1, 8 and 15
* Calaspargase 2500units/m^2/dose IV, Day 2 (Calaspargase may be replaced by alternative forms of asparaginase and will be omitted for patients in exploratory cohort N)
* Dasatinib 80mg/m^2/day PO (Max 140mg) days 1-21 for ABL-class fusions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Relapsed or refractory acute lymphoblastic leukemia or lymphoma with ≥1% bone marrow disease as measured by flow cytometry, PCR, or next generation sequencing. However, if an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the peripheral blood.
  * Patients with 1-4.99% bone marrow involvement must have disease confirmed in one of the following ways: an alternative minimal residual disease assay (e.g. flow cytometry and PCR or NGS), cytogenetic abnormality consistent with patient's leukemia, FISH abnormality, or a second bone marrow with MRD ≥1% separated by 1-4 weeks.
  * Patients with ≥5% bone marrow disease by a single measurement as measured by flow cytometry, PCR, or next generation sequencing do not require a second confirmatory test.
  * Refractory disease is defined as residual leukemia ≥1% after at least 2 prior lines of frontline therapy with curative intent.
  * Patients in exploratory cohort I must have measurable extramedullary disease but may have <1% bone marrow disease.
  * Patients in exploratory cohort M must have ≥1% bone marrow disease as measured by flow cytometry of mixed phenotype acute leukemia (MPAL)/ acute leukemia of ambiguous lineage (ALAL).
* Age ≥4 to < 30 years. Patients ≥ 22 years old are only eligible for exploratory cohort O. Sites may have different (lower) maximum ages based on institutional guidelines but may not exceed 30 years.
* Patient weighs ≥ 20 kg.
* Patient is able to swallow pills.
* Lansky/Karnofsky score is ≥ 60%. The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years.
* Participant has adequate organ function as defined by the following:

  * Direct bilirubin ≤ 1.5x the institutional upper limit of normal (ULN) unless attributable to leukemic involvement. At institutions which do not obtain a direct bilirubin in patients with a normal total bilirubin, a normal total bilirubin may be used as evidence that the direct bilirubin is not > 1.5x the ULN. Patients with a direct bilirubin ≥ 2 mg/dl may not enroll regardless of attribution.
  * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0 x the ULN unless increase is attributable to leukemic involvement.
  * Normal creatinine for age or a calculated creatinine clearance ≥ 60 mL/min/1.73 m^2.
  * Left ventricular ejection fraction (LVEF) ≥ 40% or shortening fraction ≥ 25%.

    * Patients with a history of reduced LVEF which subsequently improved with medical management are eligible if they meet the criteria above.
* Patients must have fully recovered from the acute effects of all prior therapy (defined as resolution of all such toxicities to ≤ Grade 2).
* For patients with prior hematopoietic stem cell transplant (HSCT), at least 90 days must have elapsed since transplant, the patient cannot have evidence of active graft-versus-host disease (GVHD), and they must be off calcineurin inhibitors for ≥4 weeks, and off other immunosuppression for ≥2 weeks.
* Patients with Down Syndrome/ germline Trisomy 21 are eligible for Block 1 and Block 2b therapies but are ineligible for Block 2a therapy. Patients with Down Syndrome and CD19-negative disease are off therapy after the response evaluation to Block 1.
* Prior therapy

  * ≥14 days must have elapsed since the completion of cytotoxic therapy, with the exception of standard maintenance therapy (glucocorticoids, vincristine, methotrexate, 6-mercaptopurine), tyrosine kinase inhibitors, and steroids.
  * Cytoreduction with prednisone, methylprednisolone, or hydroxyurea for ≤ 120 hours (5 days) in patients with hyperleukocytosis or extramedullary disease compromising organ function can be initiated and continued until up to 24 hours prior to the start of protocol therapy.
  * At least 21 days must have elapsed since completion of therapy with a biologic agent excluding blinatumomab. For agents that have known adverse events occurring beyond 21 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur. At least 7 days must have elapsed since blinatumomab infusion and patients must have recovered from all toxicities as described above.
  * Intrathecal cytotoxic therapy: No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone. Intrathecal chemotherapy given at the time of diagnostic LP to evaluate for relapse prior to study enrollment is allowed.
  * Patient has not had prior exposure to navitoclax
* Male or female participant of reproductive potential must agree to use appropriate methods of contraception for the duration of study treatment and for at least 30 days after last dose of protocol treatment.
* Additional criteria for exploratory cohorts

  * Cohort I: Diagnosis of isolated extramedullary relapse as defined by bone marrow blasts of <1% AND 1) central nervous system white blood cell count (WBC) of ≥ 5WBC/mL with blasts or 2) biopsy confirmed extramedullary leukemia.
  * Cohort M: Diagnosis of relapsed or refractory mixed phenotype acute leukemia (MPAL)/ acute leukemia of ambiguous lineage (ALAL).
  * Cohort N: Patients with relapsed or refractory ALL who, in the view of the provider, are unable to tolerate further asparaginase therapy due to prior toxicities.
  * Cohort O: Patients with relapsed or refractory ALL who are ages 22-29.9 years. This cohort may not enroll patients at all sites based on institutional guidelines or capacity.

Exclusion Criteria:

* Known HIV infection or active hepatitis B (defined as hepatitis B surface antigen-positive) or C (defined as hepatitis C antibody-positive).
* Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment).
* Concomitant medications and food:

  * Treatment with moderate or strong cytochrome P450 3A (CYP3A) inhibitors within 3 days of starting protocol therapy.
  * Treatment with moderate or strong CYP3A inducers within 7 days of starting protocol therapy.
  * Administration or consumption within 3 days prior to the first dose of study drug or grapefruit or grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2027-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five participants enrolled between August 25,2022 and May 3,2024. All participants initially received Block 1 therapy. Twenty-three participants completed Block 1 and met the criteria for Block 2 therapy: 7 participants enrolled on Block 2a and 16 participants enrolled on Block 2b. Ten participants only received Block 1 therapy because they did not meet the criteria for Block 2 or the treating physician recommended other therapy; two participants did not complete Block 1 because of death.
Pre-assignment Details: Participants treated on block 2a were all treated at dose level 1. Participants treated on block 2b were all treated at dose level 1.
  No participants were treated on the other dose levels.
Groups:
- Block 1: All Eligible Patients Receive Common Intervention: All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Navitoclax, Dexamethasone, Vincristine, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Dasatinib, Leucovorin, Intrathecal (IT) MHA (methotrexate/hydrocortisone/cytarabine)
  Venetoclax: Given oral (PO).
  Navitoclax: Given oral (PO).
  Dexamethasone: Given orally (PO) or intravenously (IV).
  Vincristine: Given intravenously (IV).
  Calaspargase Pegol: Given intravenously (IV).
  Dasatinib: Given oral (PO).
  Leucovorin: Given oral (PO) or intravenously (IV).
  Intrathecal Triples: Given Intrathecal (IT).
  Pegaspargase: May be used in place of Calaspargase Pegol where available. Given intravenously (IV) or intramuscularly (IM).
  Erwinia asparaginase: To be used in case of hypersensitivity or intolerance to Calaspargase Pegol or Pegaspargase. Given intravenously (IV) or intramuscularly (IM).
- Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours: Therapy for patients with ≥ 5% of leukemic blasts which do not have detectable CD19 on their surface, those with isolated extramedullary relapse, or whose physician determines this therapy arm is in their patient's best interest. All such patients completed Block 1 just prior to treatment with block 2a. These patients are mutually exclusive of patients treated on block 2b.
- Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses: Therapy for patients with>95% of leukemic blasts with detectable CD19 on their surface. All such patients completed block 1 just prior to treatment with block 2b. These patients are mutually exclusive of patients treated on block 2a.
Period: Block 1: All Eligible Patients
Arm/Group | Block 1: All Eligible Patients Receive Common Intervention | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses
Started | 35 | 0 | 0
Completed (Ten participants only received Block 1 therapy because they did not meet the criteria for Block 2 or the PI recommended other therapy.) | 33 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Death | 2 | 0 | 0
Period: Block 2a - Dose Level 1
Arm/Group | Block 1: All Eligible Patients Receive Common Intervention | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses
Started | 0 | 7 | 0
Completed | 0 | 7 (5 participants expired after completing Block 2a therapy but were still on study at the time of their deaths.) | 0
Not Completed | 0 | 0 | 0
Period: Block 2b - Dose Level 1
Arm/Group | Block 1: All Eligible Patients Receive Common Intervention | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses
Started | 0 | 0 | 16
Completed | 0 | 0 | 13 (4 participants expired after completing Block 2b therapy but were still on study at the time of their deaths.)
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Refused Therapy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Block 1: All eligible patients receive common intervention according to the Detailed Description section with the following:
  Venetoclax, Navitoclax, Dexamethasone, Vincristine, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Dasatinib, Leucovorin, Intrathecal (IT) MHA (methotrexate/hydrocortisone/cytarabine)
  Venetoclax: Given oral (PO).
  Navitoclax: Given oral (PO).
  Dexamethasone: Given orally (PO) or intravenously (IV).
  Vincristine: Given intravenously (IV).
  Calaspargase Pegol: Given intravenously (IV).
  Dasatinib: Given oral (PO).
  Leucovorin: Given oral (PO) or intravenously (IV).
  Intrathecal Triples: Given Intrathecal (IT).
  Pegaspargase: May be used in place of Calaspargase Pegol where available. Given intravenously (IV) or intramuscularly (IM).
  Erwinia asparaginase: To be used in case of hypersensitivity or intolerance to Calaspargase Pegol or Pegaspargase. Given intravenously (IV) or intramuscularly (IM).
Arm/Group | Block 1
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.99 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22
  Black | 6
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Minimal Residual Disease (MRD)-Negative Response
Description: The number of participants with end Block 1 minimal residual disease <0.01% by flow cytometry
Time Frame: 4 weeks from start of therapy
Population: Of the 35 patients, 30 Patients had MRD data at the end of Block 1, and 5 patients with no adequate sample.
Measure: Count of Participants; unit: Participants
Groups:
- Block 1: All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Navitoclax, Dexamethasone, Vincristine, Calaspargase Pegol, Pegaspargase, Erwinia asparaginase, Dasatinib, Leucovorin, Intrathecal (IT) MHA (methotrexate/hydrocortisone/cytarabine)
  Venetoclax: Given oral (PO).
  Navitoclax: Given oral (PO).
  Dexamethasone: Given orally (PO) or intravenously (IV).
  Vincristine: Given intravenously (IV).
  Calaspargase Pegol: Given intravenously (IV).
  Dasatinib: Given oral (PO).
  Leucovorin: Given oral (PO) or intravenously (IV).
  Intrathecal Triples: Given Intrathecal (IT).
  Pegaspargase: May be used in place of Calaspargase Pegol where available. Given intravenously (IV) or intramuscularly (IM).
  Erwinia asparaginase: To be used in case of hypersensitivity or intolerance to Calaspargase Pegol or Pegaspargase. Given intravenously (IV) or intramuscularly (IM).
Arm/Group | Block 1
Number analyzed (Participants) | 30
Participants | 19

2. Primary Outcome: Recommended Phase 2 Dose of Venetoclax in Combination With a) High-dose Cytarabine and Navitoclax
Description: The recommended Phase 2 dose (RP2D) of venetoclax in combination with a) high-dose cytarabine and navitoclax will be the dose at which 0 or 1 of 6 treated patients experience a dose limiting toxicity.
Time Frame: 6 weeks from the start of block 2a
Population: Participants treated at Dose Level 1 in Block 2a during dose finding.
Measure: Number; unit: mg/m^2 for cytarabine
Groups:
- Block 2: Includes participants treated with Block 2a therapy.
Arm/Group | Block 2
Number analyzed (Participants) | 6
mg/m^2 for cytarabine | 3000

3. Primary Outcome: Recommended Phase 2 Dose of Venetoclax in Combination With b) Blinatumomab
Description: The recommended Phase 2 dose (RP2D) of venetoclax in combination with b) blinatumomab will be the dose at which 0 or 1 of 6 treated patients experience a dose limiting toxicity. RP2D is 240mg/m2 which was delivered for 21 days.
Time Frame: 4 weeks from the start of block 2b
Population: Participants treated at Dose Level 1 in Block 2b during dose finding.
Measure: Number; unit: 240 mg/m^2/day
Groups:
- Block 2b: Includes participants treated with Block 2b therapy.
Arm/Group | Block 2b
Number analyzed (Participants) | 6
240 mg/m^2/day | 240

4. Secondary Outcome: Number of Participants With Grade 3 or Higher CTCAE Events in Block 2a
Description: Occurrence of grade 3 or higher CTCAE version 5 events in patients receiving block 2a therapy estimated as a proportion of patients receiving that therapy
Time Frame: 6 weeks from start of block 2a
Population: Among the 7 patients who went to block 2a, 6 of them had Grade>=3 CTCAE version 5 events.
Measure: Count of Participants; unit: Participants
Groups:
- Block 2a: Includes participants treated with Block 2a therapy.
Arm/Group | Block 2a
Number analyzed (Participants) | 7
Participants | 6

5. Secondary Outcome: Number of Participants With Grade 3 or Higher CTCAE Events in Block 2b
Description: Occurrence of grade 3 or higher CTCAE version 5 events in patients receiving block 2b therapy estimated as a proportion of patients receiving that therapy
Time Frame: 4 weeks from start of block 2b
Population: Among the 16 patients who went to block 2b, 3 of them had Grade>=3 CTCAE version 5 events.
Measure: Count of Participants; unit: Participants
Arm/Group | Block 2b
Number analyzed (Participants) | 16
Participants | 3

6. Secondary Outcome: Event Free Survival (EFS)
Description: EFS will be reported as estimates using the Kaplan-Meier method
Time Frame: 1, 3 and 5 years from study entry
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OS)
Description: OS will be reported as estimates using the Kaplan-Meier method
Time Frame: 1, 3 and 5 years from study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants will be followed for adverse events from the time the of signed study specific informed consent/assent throughout the time of study drug administration until 30 days following discontinuation of study drug administration, up to 3 years.
Groups:
- Block 1: All patients receive common therapy.
- Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours: Therapy for patients with ≥ 5% of leukemic blasts which do not have detectable CD19 on their surface, those with isolated extramedullary relapse, or whose physician determines this therapy arm is in their patient's best interest.
- Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses: Therapy for patients with >95% of leukemic blasts with detectable CD19 on their surface.
- Post Therapy Follow-up: Follow-up after completion of protocol therapy. This is inclusive of all patients treated with block 1 therapy including those who did and did not proceed to block 2a or 2b therapy. Such description enables understanding of the during vs. post therapy toxicity experienced by participants.
Arm/Group | Block 1 | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses | Post Therapy Follow-up
All-Cause Mortality (participants affected / at risk) | 2/35 | 0/7 | 0/16 | 16/33
Serious Adverse Events (participants affected / at risk) | 8/35 | 2/7 | 0/16 | 0/33
Other Adverse Events (participants affected / at risk) | 15/35 | 1/7 | 2/16 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Block 1 (N=35) | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours (N=7) | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses (N=16) | Post Therapy Follow-up (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 2 | 0 | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | NA
Typhlitis (Gastrointestinal disorders) | 2 | 1 | 0 | NA
Appendicitis (Infections and infestations) | 1 | 0 | 0 | NA
Infections and infestations - Other, specify (Infections and infestations) | 8 | 0 | 0 | NA
Lung infection (Infections and infestations) | 0 | 1 | 0 | NA
Meningitis (Infections and infestations) | 1 | 0 | 0 | NA
Sepsis (Infections and infestations) | 5 | 0 | 0 | NA
Shingles (Infections and infestations) | 0 | 1 | 0 | NA
Sinusitis (Infections and infestations) | 1 | 0 | 0 | NA
Skin infection (Infections and infestations) | 1 | 0 | 0 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA
Seizure (Nervous system disorders) | 1 | 0 | 0 | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | NA
Confusion (Psychiatric disorders) | 1 | 0 | 0 | NA
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Block 1 (N=35) | Block 2a - Dose Level 1: Cytarabine 3000mg/m^2/Dose Every 12 Hours (N=7) | Block 2b - Dose Level 1: Venetoclax 240mg/m^2 for 21 Doses (N=16) | Post Therapy Follow-up (N=33)
Aspartate aminotransferase increased (Investigations) | 15 | 0 | 0 | NA
Alanine aminotransferase increased (Investigations) | 11 | 1 | 1 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 0 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 11 | 0 | 0 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 0 | 0 | NA
Infections and infestations - Other, specify (Infections and infestations) | 6 | 0 | 0 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA
Sepsis (Infections and infestations) | 2 | 0 | 0 | NA
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | NA
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Ascites (Investigations) | 1 | 0 | 0 | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Bacteremia (Infections and infestations) | 1 | 0 | 0 | NA
Blood bilirubin increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Blurred vision (Eye disorders) | 1 | 0 | 0 | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0 | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 | 0 | 0 | NA
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Headache (Nervous system disorders) | 1 | 0 | 1 | NA
Herpes simplex reactivation (Infections and infestations) | 1 | 0 | 0 | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hypertension (Vascular disorders) | 1 | 0 | 0 | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Lipase increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA
Peripheral sensory neuropathy (Vascular disorders) | 1 | 0 | 0 | NA
Shingles (Infections and infestations) | 1 | 0 | 0 | NA
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | NA
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | NA
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 | NA
Sinusitis (Infections and infestations) | 0 | 1 | 0 | NA
Skin infection (Infections and infestations) | 0 | 0 | 2 | NA
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | NA
Pruritus (Infections and infestations) | 0 | 0 | 1 | NA
Seizure (Nervous system disorders) | 0 | 0 | 1 | NA
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT05192889/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT05192889/ICF_000.pdf